CLINICAL TRIAL: NCT02460029
Title: Prospective MRI Follow-up After Retromuscular Incisional Hernia Repair Using the Dynamesh CICAT Visible® Mesh
Brief Title: MRI Imaging of Retromuscular Hernia Repair With CICAT Visible®
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Collaborators: Duomed (Industry)
Responsible Party: Principal Investigator, Filip Muysoms, Head of the Department of Surgery, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: MoonCat Study
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hernia; Recurrence
MeSH Terms: conditions — Hernia; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Other: Ventral hernia — Visualization of the mesh surface and the confirmation with MRI scan at 1 month and 13 months after standardized retromusculare incisional hernia repair with the visible CICAT mesh (Dynamesh®).

SUMMARY:
The aim of this study is the visualization of the mesh surface and the confirmation with MRI scan at 1 month and 13 months after standardized retromuscular incisional hernia repair with the visible CICAT mesh (Dynamesh®).

DETAILED DESCRIPTION:
INTRODUCTION:

Repair of ventral hernias always involves a scientific discussion about placing the "optimal mesh", the "optimal" mesh position or the "optimal" fixation method of the mesh. Today, there are a lot of meshes available of different materials, different textures, in different sizes and with different properties. The choice of the "right" mesh strongly depends on the sort of hernia and on the choice of the surgeon.

Furthermore, it is known that the majority of implanted meshes shrink to an extent, which may be of disadvantage for the patient. This has already been demonstrated in several animal studies, but clinical information on the mesh shrinkage is rare and mostly a result from revised surgery.

Most meshes for repair of abdominal hernia defects, based on polymeric textile, are invisible to conventional imaging techniques, inclusive "magnetic resonance imaging" (MRI). The textile company FEG Textiltechnik GmbH, Germany, has developed a unique method which allows imaging of the mesh in vivo in the MRI. For this purpose, these unique meshes contain an amount of iron particles. The particles are incorporated into the filaments, which are subsequent warp knitted to the mesh structure.

In a similar setting, the IMAP study, the visibility of the IPOM® mesh up to 13 months after laparoscopic ventral hernia repair will be investigated. Preliminary results from this study have shown a clear visibility and a promising outcome using this mesh.

PURPOSE:

The aim of this study is the visualization of the mesh surface and the confirmation with MRI scan at 1 month and 13 months after standardized retromuscular incisional hernia repair with the visible CICAT mesh (Dynamesh®).

The investigators want to show that with this type of mesh it is possible to visualize the mesh after retromuscular placement in vivo in a safe manner.

Furthermore, the positioning of the mesh, mesh shrinkage or mesh shifting will be monitored with this technique. This provides long-term benefit and provides early treatment possibilities in case of post-operative complications related to the mesh position. Furthermore, by means of dynamic MRI measurements the mesh elasticity will be evaluated in both directions longitudinal as well as transversal.

These results will provide information about the degree of mesh incorporation and the mechanical behavior of the tissue-mesh compound.

PROCEDURES

Hernia Repair:

* Introduction of the visible CICAT mesh (Dynamesh®) via laparotomy and retromuscular positioning of the mesh with a minimum overlap with the hernia defect of at least 5 cm in all directions.
* All patients will receive a standardized pain treatment protocol. Analgesics used will be checked. Visual analog scale (VAS) for pain will be measured at 4 hours, 8 hours, 12 hours, 16 hours, 20 hours and 24 hours post-operatively and every 12 hours thereafter until discharge of the patient.
* Pain medication after discharge will be monitored and checked with the patient at each consultation.

Clinical follow-up evaluation of all patients will be performed by the principal investigator.

MRI measurement will be performed at 1 and 13 months post-operatively.

MRI scan method:

Used gear: Philips Ingenia CX 1.5 Tesla. Measurements will be performed in head first prone position and if not possible in head first supine position. Prone position is preferred because of less motion artefacts from respiration and aortic pulsation, less tendency of intestinal gas accumulation against the abdominal wall producing additional signal voids. Hence the differentiation with the hypointense mesh can be difficult.

There is no use of contrast material during the investigation. Preferably, the examination will be conducted in sober state i.e. patient should not eat for 2 hours before the examination. This is to reduce the risk of post prandial hyper-peristaltic.

DATA PROTECTION AND PRIVACY OF THE PATIENT All information about this study will be collected in the EuraHS Registry. The data will be entered into the EuraHS platform with a coded number, MOONCAT_01, MOONCAT_02, ...

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for an retromusculare repair of an incisional hernia

Exclusion Criteria:

* <18 years
* Emergency surgery (incarcerated hernia)
* Clean-contaminated or contaminated procedures
* ASA score> 4
* Pregnancy
* No patient Informed Consent
* Life expectancy of less than 2 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for an open retromusculare repair of an incisional hernia.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-05; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
visualization of the mesh surface | 1 month
  Clear visualization of the CICAT® prosthesis at 1 month postoperatively with MRI

SECONDARY OUTCOMES:
calculation of the mesh surface | up to 13 months
  Calculation of mesh surface in comparison and % difference at 13 months postoperatively with MRI.
visualization of the mesh surface | up to 13 months
  Clear visualization of the CICAT® prosthesis up to 13 months postoperatively with MRI

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD. PhD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen NL, Ciritsis A, Otto J, Busch D, Kuhl CK, Kraemer NA. Utility of Magnetic Resonance Imaging to Monitor Surgical Meshes: Correlating Imaging and Clinical Outcome of Patients Undergoing Inguinal Hernia Repair. Invest Radiol. 2015 Jul;50(7):436-42. doi: 10.1097/RLI.0000000000000148. PMID 25756683
- [Result] Ciritsis A, Hansen NL, Barabasch A, Kuehnert N, Otto J, Conze J, Klinge U, Kuhl CK, Kraemer NA. Time-dependent changes of magnetic resonance imaging-visible mesh implants in patients. Invest Radiol. 2014 Jul;49(7):439-44. doi: 10.1097/RLI.0000000000000051. PMID 24651663
- [Result] Hansen NL, Barabasch A, Distelmaier M, Ciritsis A, Kuehnert N, Otto J, Conze J, Klinge U, Hilgers RD, Kuhl CK, Kraemer NA. First in-human magnetic resonance visualization of surgical mesh implants for inguinal hernia treatment. Invest Radiol. 2013 Nov;48(11):770-8. doi: 10.1097/RLI.0b013e31829806ce. PMID 23732864